CLINICAL TRIAL: NCT02350140
Title: Texting to Improve Testing (TextIT): A Cluster Randomized Stepped Wedge Trial of Text Messaging to Improve Postpartum Retention in Care and Early Infant Diagnosis of HIV
Brief Title: Texting to Improve Testing (TextIT):
Acronym: TextIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas Odeny, Research Scientist, Kenya Medical Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 41186
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2017-11

CONDITIONS: HIV
Keywords: HIV; Prevention of mother-to-child HIV transmission; PMTCT; mobile health (mHealth); mobile phone; text messaging; short message services (SMS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text messaging from beginning (Experimental): Half of the health facilities will be randomly allocated to receive the TextIT intervention during the first time period (six months), while the other half to continue with current standard care (first step)
  Interventions: Other: Text messaging from beginning
- Text messaging after 6 months of control (Active Comparator): Half the facilities will receive standard of care for six months (first time period). After the first time period, the these facilities will then also receive the TextIT intervention (second step)
  Interventions: Other: Text messaging after 6 months of control

INTERVENTIONS:
Other: Text messaging from beginning — Registered women will then receive up to 14 text messages as follows: weeks 28, 30, 32, 34, 36, 38, 39, and 40 during the third trimester of pregnancy; weeks 1, 2, 3, 4, 5, and 6 after delivery.Participants at facilities receiving TextIT will have the option to call or send text messages to a designated clinic phone, to which a clinic nurse will respond. Participants will also have an option to request a call from the clinic by sending a free "call back" text message to the designated clinic phone at any time.
  Other Names: TextIT
  Arms: Text messaging from beginning
Other: Text messaging after 6 months of control — After six months of standard care, women at control clinics will be registered to receive the text messaging intervention with up to 14 text messages as follows: weeks 28, 30, 32, 34, 36, 38, 39, and 40 during the third trimester of pregnancy; weeks 1, 2, 3, 4, 5, and 6 after delivery.
  Arms: Text messaging after 6 months of control

SUMMARY:
Early accurate diagnosis is one of the first crucial steps in care for infants born to HIV-infected mothers. Early initiation of antiretroviral therapy (ART) relies upon early diagnosis and results in significant reductions in infant morbidity and mortality. The investigators recently concluded a successful randomized controlled trial in Kenya entitled, "Improving uptake of early infant diagnosis of HIV for prevention of mother-to-child HIV transmission (PMTCT): a randomized trial of a text messaging intervention" (ClinicalTrials.gov # NCT01433185). In this study, text messages developed using a behavioral theoretical framework significantly improved maternal attendance at post-partum clinic appointments and rates of testing to facilitate early infant diagnosis of HIV in a selected population and controlled setting. Understanding the effectiveness of this intervention (and its limitations) in a real-world, routine-care setting represents the next step in the translational pathway to public health impact. The investigators therefore now propose a cluster randomized, stepped wedge trial in 20 clinics operated by the Kenyan Ministry of Health in the Nyanza region of Kenya and use the Reach, Effectiveness, Adoption, Implementation, and Maintenance (REAIM) framework to understand the effectiveness of the text messaging to improve testing (TextIT) intervention. Our specific aims are:

1. To determine the effect of TextIT on maternal attendance at postpartum clinic visits during the randomized stepped-wedge rollout of the intervention.

   Hypothesis 1: A greater proportion of women at health facilities implementing TextIT will attend clinic within eight weeks postpartum compared to women at health facilities implementing standard care.
2. To determine the effect of TextIT on virological infant HIV testing within eight weeks after birth during the randomized stepped-wedge rollout of the intervention.

   Hypothesis 2: Infants of women at health facilities implementing TextIT will be more likely to have virological HIV testing compared to infants of women at health facilities implementing standard care.
3. To determine the costs and cost-effectiveness of TextIT. The investigators will estimate the cost per patient and per health gain achieved (disability-adjusted life year, DALY) comparing TextIT to current standard care.

Hypothesis 3: The TextIT intervention will be more cost-effective than current standard care.

DETAILED DESCRIPTION:
The 2011 United Nations General Assembly Political Declaration on HIV/AIDS set a target to eliminate mother-to-child transmission of HIV by 2015. The continuum of care for women living with HIV and their babies includes retention in care and early infant diagnosis of HIV. Timely initiation of infant antiretroviral therapy (ART) requires HIV-positive women to be retained in care through the postpartum period and to bring their children for HIV testing. However, a high proportion of pregnant HIV-positive women in sub-Saharan Africa are lost to follow-up after delivery. The World Health Organization recommends infant HIV testing at six weeks using DNA polymerase chain reaction (PCR). However, the overall proportion of children who undergo early infant diagnosis by PCR remains low. In Kenya, the overall proportion of eligible children undergoing PCR testing in 2011 was 39%.

Low rates of infant HIV testing are an indirect indication of a large number of infants who may not benefit from early determination of HIV status, antiretroviral prophylaxis for HIV-negative breastfeeding infants, and infant feeding counseling and support. For HIV positive infants, failure to undergo testing is a critical barrier to receiving life-saving ART. There is an urgent need to investigate efficacious, cost-effective, and sustainable interventions to improve maternal retention in HIV care and increase the proportion of exposed infants tested for HIV.

With the exponential increase in the number of mobile phones in sub-Saharan Africa, the use of mobile technology to support HIV programs has shown promise. The United Nations Children's Fund is encouraging HIV programs to take advantage of high levels of mobile phone access among enrolled mothers by reminding them to return for critical appointments. Active follow-up of pregnant HIV positive women in resource-limited settings using mobile phones is feasible, and may be effective in improving postnatal retention and uptake of early infant diagnosis across different sub-Saharan African settings.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥18 years or emancipated minors;
* Are at 28 weeks gestation or greater (or have delivered on the day of enrollment);
* Provide informed consent

Exclusion Criteria:

* Women who report sharing phones but have not disclosed their HIV status to the person with whom the phone is shared.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2508 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum retention in prevention of mother-to-child HIV transmission programs | 1 year
  Maternal attendance at postpartum clinic visits within eight weeks after delivery
Infant HIV testing by DNA PCR within 8 weeks after birth | 1 year
Cost-effectiveness of TextIT | 1 year

SECONDARY OUTCOMES:
Overall public health impact | 1 year
  To determine the overall public health impact of the TextIT strategy using the REAIM framework which assesses five dimensions of public health interventions: Reach, Effectiveness, Adoption, Implementation, and Maintenance
Place of delivery and skilled birth attendance | 1 year
A combined outcome for stillbirth (after 28 weeks of pregnancy) or infant death within the first two months after a live birth | 1 year
Birth weight | 1 year
Reported infant feeding option | 1 year
Incidence rate of HIV-1 among infants who undergo virological HIV testing | 1 year
18 month PMTCT outcomes | 18 months
  Includes discharge from the PMTCT program, referral and linkage to the general HIV comprehensive care clinic, transfer out to another health facility, lost to follow-up or death; and infant HIV status by antibody testing.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Odeny, MBChB, MPH, Principal Investigator — Kenya Medical Research Institute; Scott R McClelland, MD MPH, Study Chair — University of Washington; Craig R Cohen, MD MPH, Study Chair — University of California, San Francisco; Elizabeth Bukusi, MBCHB PHD, Study Chair — Kenya Medical Research Institute
Locations (1):
- Kenya Medical Research Institute, Family AIDS Care and Education Services, Kisumu, Nyanza, Kenya

REFERENCES:
- [Background] Odeny TA, Bukusi EA, Cohen CR, Yuhas K, Camlin CS, McClelland RS. Texting improves testing: a randomized trial of two-way SMS to increase postpartum prevention of mother-to-child transmission retention and infant HIV testing. AIDS. 2014 Sep 24;28(15):2307-12. doi: 10.1097/QAD.0000000000000409. PMID 25313586
- [Background] Odeny TA, Newman M, Bukusi EA, McClelland RS, Cohen CR, Camlin CS. Developing content for a mHealth intervention to promote postpartum retention in prevention of mother-to-child HIV transmission programs and early infant diagnosis of HIV: a qualitative study. PLoS One. 2014 Sep 2;9(9):e106383. doi: 10.1371/journal.pone.0106383. eCollection 2014. PMID 25181408
- [Derived] Odeny TA, Hughes JP, Bukusi EA, Akama E, Geng EH, Holmes KK, McClelland RS. Text messaging for maternal and infant retention in prevention of mother-to-child HIV transmission services: A pragmatic stepped-wedge cluster-randomized trial in Kenya. PLoS Med. 2019 Oct 2;16(10):e1002924. doi: 10.1371/journal.pmed.1002924. eCollection 2019 Oct. PMID 31577792